CLINICAL TRIAL: NCT02992925
Title: Phase 3 Study of BK1310 in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: The Research Foundation for Microbial Diseases of Osaka University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BK1310-J01
Record Dates: First submitted 2016-12-01; First posted 2016-12-14 (Estimated); Results first posted 2025-01-07 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Immunization; Infection
Keywords: Haemophilus influenza type b; Adsorbed Diphteria-purified Pertussis-Tetanus-Inactivate poliovirus combined vaccine; Hib; DPT-IPV
MeSH Terms: conditions — Infections; Haemophilus Infections | interventions — HibTITER protein, Haemophilus influenzae; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1: BK1310-High (Experimental)
  Interventions: Biological: DPT-IPV-Hib-High（Combined Vaccine）
- Cohort 1: BK1310-Low (Experimental)
  Interventions: Biological: DPT-IPV-Hib-Low（Combined Vaccine）
- Cohort 2: BK1310-High or -Low (Experimental): Either BK1310-High or -Low will be chosen based on the result of cohort 1
  Interventions: Biological: DPT-IPV-Hib-High（Combined Vaccine）; Biological: DPT-IPV-Hib-Low（Combined Vaccine）
- Cohort 2: ActHIB® and Tetrabik (Active Comparator)
  Interventions: Biological: Hib vaccine; Biological: DPT-IPV

INTERVENTIONS:
Biological: DPT-IPV-Hib-High（Combined Vaccine）
  Other Names: BK1310-High
  Arms: Cohort 1: BK1310-High; Cohort 2: BK1310-High or -Low
Biological: DPT-IPV-Hib-Low（Combined Vaccine）
  Other Names: BK1310-Low
  Arms: Cohort 1: BK1310-Low; Cohort 2: BK1310-High or -Low
Biological: Hib vaccine
  Other Names: ActHIB®
  Arms: Cohort 2: ActHIB® and Tetrabik
Biological: DPT-IPV
  Other Names: Tetrabik
  Arms: Cohort 2: ActHIB® and Tetrabik

SUMMARY:
The purpose of this study is to:

* (cohort 1) evaluate safety and immunogenicity (Haemophilus influenzae type b, Hib) of BK1310.
* (cohort 2) evaluate efficacy and safety of BK1310 using ActHIB® and Tetrabik as a control in healthy infants.

DETAILED DESCRIPTION:
<Cohort 1>

* Arm: BK1310-High. Intervention: DPT-IPV-Hib-High(Combined Vaccine) 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.
* Arm: BK1310-Low. Intervention: DPT-IPV-Hib-Low(Combined Vaccine) 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.

<Cohort 2>

* Arm: BK1310-High or Low. Intervention: DPT-IPV-Hib-High(Combined Vaccine) or DPT-IPV-Hib-Low(Combined Vaccine) 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals.
* Arm: ActHIB® and Tetrabik. Intervention: Hib vaccine and DPT-IPV 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged ≥2 and <43 months at the first vaccination of the study drug (recommended: ≥2 and <7 months). Those who are applicable of the following conditions must be carefully observed before the enrollment: infants with known underlying disease such as cardiovascular disease, renal disease, hepatic disease, blood dyscrasia, respiratory disease or developmental disorder. Infants who developed fever within 2 days after any previous vaccination. Infants with history of convulsions.
* Written informed consent is obtained from a legal guardian (parent)

Exclusion Criteria:

* With past diagnosis of immunodeficiency or currently under immunosuppressive treatment
* Have close relatives (the third degree of kinship) diagnosed with congenital immunodeficiency
* Possibility of anaphylaxis due to food or pharmaceuticals
* With experience of Hib infection, diphtheria, pertussis, tetanus or acute poliomyelitis
* With experience of Hib, diphteria, pertussis, tetanus or polio vaccination.
* Administered a live vaccine within 27 days before the first vaccination of the study drug, or inactivated vaccine or toxoid within 6 days before vaccination
* Administered transfusion, immunosuppressant (excluding drugs for external use), or immunoglobulin formulation
* Administered corticosteroid 2 mg/kg per day or more as prednisolone (excluding drugs for external use)
* Participated in other studies within 12 weeks before obtaining consent
* With the gestational age <37 weeks or weighed less than 2500 grams at birth.
* Considered to be not eligible by the principal investigators (sub-investigators) of the enrollment.

Ages: 2 Months to 43 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 370 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (3):
- Japan (3):
  - Fukuoka, Fukuoka
  - Kasuga-shi, Fukuoka
  - Sendai, Miyagi

RESULTS

PARTICIPANT FLOW:
Groups:
- BK1310-High: (Cohort 1) DPT-IPV-Hib-High(Combined Vaccine) 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.
- BK1310-Low: (Cohort 1) DPT-IPV-Hib-Low(Combined Vaccine) 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.
- BK1310: (Cohort 2) DPT-IPV-Hib-High(Combined Vaccine) 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals.
- ActHIB® and Tetrabik (Control): (Cohort 2) Hib vaccine and DPT-IPV 0.5mL, subcutaneous injection, 3 times with the 3-8weeks intervals.
Period: Cohort 1
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Started | 15 (15 subjects of BK1310-High group were finished in cohort 1.) | 15 (15 subjects of BK1310-Low group were finished in cohort 1.) | 0 (171 subjects of BK1310 group were started from cohort 2.) | 0 (169 subjects of BK1310 group were started from cohort 2.)
Completed | 15 | 15 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Started | 0 (15 subjects of BK1310-High group were finished in cohort 1.) | 0 (15 subjects of BK1310-Low group were finished in cohort 1.) | 171 (171 subjects of BK1310 group were started from cohort 2.) | 169 (169 subjects of BK1310 group were started from cohort 2.)
Completed | 0 | 0 | 170 | 167
Not Completed | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 【cohort 2_Age,Sex/Gender】 Excluding 5 subjects(BK1310: 1 subject, control: 4 subjects) whose all antibody titers could not be measured at Visit 4
Groups:
- Total: Total of all reporting groups
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control) | Total
Number analyzed (Participants) | 15 | 15 | 170 | 165 | 365
Age, Customized [Count of Participants; unit: Participants]
  >=2 and <3 months | 7 | 6 | 154 | 145 | 312
  >=3 months | 8 | 9 | 16 | 20 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 86 | 79 | 181
  Male | 7 | 7 | 84 | 86 | 184
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 15 | 15 | 170 | 165 | 365

OUTCOME MEASURES:

1. Primary Outcome: Antibody Prevalence Rate Against Anti-PRP With 1 μg/mL or Higher, Diphtheria Toxin, Pertussis, Tetanus Toxin, and Polio Virus, Defined as the Percentage of Participants With the Antibody Against Anti-PRP
Description: Antibody prevalence rate is defined as the percentage of participants whose criteria of each antibody titer: Anti-diphtheria antibody concentrations: >=0.1 IU/mL, Anti-PT antibody concentrations: >=10.0 EU/mL, Anti-FHA antibody concentrations: >=10.0 EU/mL, Anti-tetanus antibody concentrations: >=0.01 IU/mL, Anti-poliovirus serotype 1, 2 and 3, antibody titers (fold) >=8
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects decreased from 370 to 365. BK1310 group: due to physician decision (n=1).Control group: due to withdrawal by parent/guardian (n=2) and deviation in blood collection timing (n=2). In control group number of subjects further decreased due to insufficient sample volume (diphtheria: n=2, PT: n=1, FHA: n=1, tetanus: n=1, polio serotype1: n=5, polio serotype2: n=4, polio serotype3: n=4）
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 15 | 15 | 170 | 165
percentage of participants
  Antibody prevalence rate against anti-PRP with 1 μg/mL or higher | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [97.9 to 100.0] | 93.3 [88.4 to 96.6]
  Antibody prevalence rate against diphtheria toxin: number analyzed (Participants) | 15 | 15 | 170 | 163
  Antibody prevalence rate against diphtheria toxin | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0] | 97.6 [94.1 to 99.4] | 98.8 [95.6 to 99.9]
  Antibody prevalence rate against pertussis （PT）: number analyzed (Participants) | 15 | 15 | 170 | 164
  Antibody prevalence rate against pertussis （PT） | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0] | 99.4 [96.8 to 100.0] | 100.0 [97.8 to 100.0]
  Antibody prevalence rate against pertussis (FHA): number analyzed (Participants) | 15 | 15 | 170 | 164
  Antibody prevalence rate against pertussis (FHA) | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0] | 97.6 [94.1 to 99.4] | 99.4 [96.6 to 100.0]
  Antibody prevalence rate against tetanus toxin: number analyzed (Participants) | 15 | 15 | 170 | 164
  Antibody prevalence rate against tetanus toxin | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [97.9 to 100.0] | 100.0 [97.8 to 100.0]
  Antibody prevalence rate against polio virus serotype 1: number analyzed (Participants) | 15 | 15 | 170 | 160
  Antibody prevalence rate against polio virus serotype 1 | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [97.9 to 100.0] | 100.0 [97.7 to 100.0]
  Antibody prevalence rate against polio virus serotype 2: number analyzed (Participants) | 15 | 15 | 170 | 161
  Antibody prevalence rate against polio virus serotype 2 | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [97.9 to 100.0] | 100.0 [97.7 to 100.0]
  Antibody prevalence rate against polio virus serotype 3: number analyzed (Participants) | 15 | 15 | 170 | 161
  Antibody prevalence rate against polio virus serotype 3 | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [97.9 to 100.0] | 100.0 [97.7 to 100.0]

2. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 0.15 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects decreased from 370 to 365. BK1310 group: due to physician decision (n=1).Control group: due to withdrawal by parent/guardian (n=2) and deviation in blood collection timing (n=2).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 15 | 15 | 170 | 165
percentage of participants | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [97.9 to 100.0] | 100.0 [97.8 to 100.0]

3. Secondary Outcome: Geometric Mean Antibody Titer of Anti-PRP Antibody
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 15 | 15 | 170 | 165
µg/mL | 17.613 [10.911 to 28.432] | 23.097 [14.545 to 36.680] | 17.832 [15.251 to 20.850] | 6.245 [5.177 to 7.533]

4. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 1 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: Only subjects in cohort 1 were analyzed. Visit 6 was not conducted in Cohort 2（Arm；BK-1310，ActHIB® and Tetrabik）, and the data of Cohort 2 were not collected. Therefore, no data of Cohort 2 are available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310-High | BK1310-Low
Number analyzed (Participants) | 15 | 15
percentage of participants | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0]

5. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 0.15 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310-High | BK1310-Low
Number analyzed (Participants) | 15 | 15
percentage of participants | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0]

6. Secondary Outcome: Geometric Mean Antibody Titer of Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | BK1310-High | BK1310-Low
Number analyzed (Participants) | 15 | 15
µg/mL | 69.937 [46.971 to 104.132] | 54.333 [33.441 to 88.276]

7. Secondary Outcome: Geometric Mean Antibody Titer Against Diphtheria Toxin
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects decreased from 370 to 365. BK1310 group: due to physician decision (n=1).Control group: due to withdrawal by parent/guardian (n=2) and deviation in blood collection timing (n=2). In control group number of subjects further decreased due to insufficient sample volume (diphtheria: n=2）
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 15 | 15 | 170 | 163
IU/mL | 1.1640 [0.7205 to 1.8806] | 0.8058 [0.4842 to 1.3411] | 0.8767 [0.7484 to 1.0269] | 0.7010 [0.6000 to 0.8189]

8. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis （PT）
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects decreased from 370 to 365. BK1310 group: due to physician decision (n=1).Control group: due to withdrawal by parent/guardian (n=2) and deviation in blood collection timing (n=2). In control group number of subjects further decreased due to insufficient sample volume (PT: n=1）
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 15 | 15 | 170 | 164
EU/mL | 208.80 [161.19 to 270.48] | 180.78 [114.40 to 285.69] | 175.35 [158.60 to 193.87] | 184.17 [169.75 to 199.82]

9. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis （FHA）
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects decreased from 370 to 365. BK1310 group: due to physician decision (n=1).Control group: due to withdrawal by parent/guardian (n=2) and deviation in blood collection timing (n=2). In control group number of subjects further decreased due to insufficient sample volume (FHA: n=1）
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 15 | 15 | 170 | 164
EU/mL | 67.41 [48.46 to 93.77] | 49.99 [35.86 to 69.69] | 57.59 [51.87 to 63.93] | 83.64 [75.81 to 92.28]

10. Secondary Outcome: Geometric Mean Antibody Titer Against Tetanus Toxin
Time Frame: 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects decreased from 370 to 365. BK1310 group: due to physician decision (n=1).Control group: due to withdrawal by parent/guardian (n=2) and deviation in blood collection timing (n=2). In control group number of subjects further decreased due to insufficient sample volume (tetanus: n=1）
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 15 | 15 | 170 | 164
IU/mL | 0.5320 [0.2901 to 0.9755] | 0.4032 [0.2406 to 0.6757] | 0.4950 [0.4305 to 0.5693] | 0.2807 [0.2261 to 0.3485]

11. Secondary Outcome: Fold Change in Geometric Mean Antibody Titer Against Polio Virus
Time Frame: Baseline and 4 weeks after the primary immunization (Visit 4)
Population: For antibody analysis at Visit 4, number of subjects decreased from 370 to 361. BK1310 group: due to physician decision (n=1). Control group: due to withdrawal by parent/guardian (n=2), deviation in blood collection timing (n=2), insufficient sample volume (n=4). In control group number of subjects further decreased due to insufficient sample volume (polio serotype1: n=1）
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
Number analyzed (Participants) | 15 | 15 | 170 | 161
fold change
  Geometric mean antibody titer against polio virus serotype 1: number analyzed (Participants) | 15 | 15 | 170 | 160
  Geometric mean antibody titer against polio virus serotype 1 | 933.60 [350.43 to 2487.27] | 588.13 [282.89 to 1222.76] | 742.01 [579.83 to 949.55] | 885.67 [698.16 to 1123.54]
  Geometric mean antibody titer against polio virus serotype 2 | 1824.56 [1369.18 to 2431.40] | 1955.52 [1403.94 to 2723.79] | 2137.58 [1871.07 to 2442.06] | 1978.66 [1681.86 to 2327.85]
  Geometric mean antibody titer against polio virus serotype 3 | 851.19 [494.94 to 1463.86] | 1320.32 [813.95 to 2141.70] | 1430.55 [1230.96 to 1662.49] | 1551.43 [1339.55 to 1796.81]

12. Secondary Outcome: Antibody Prevalence Rate Against Diphtheria Toxin, Pertussis, Tetanus Toxin, and Polio Virus, Defined as the Percentage of Participants With the Antibody Against Diphtheria Toxin, Pertussis, Tetanus Toxin, and Polio Virus
Description: Antibody prevalence rate is defined as the percentage of participants whose criteria of each antibody titer: Anti-diphtheria antibody concentrations: >=0.1 IU/mL, Anti-PT antibody concentrations: >=10.0 EU/mL, Anti-FHA antibody concentrations: >=10.0 EU/mL, Anti-tetanus antibody concentrations: >=0.01 IU/mL, Anti-poliovirus serotype 1,2 and 3 antibody titers (fold) >=8
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310-High | BK1310-Low
Number analyzed (Participants) | 15 | 15
percentage of participants
  Antibody prevalence rate against diphtheria toxin | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0]
  Antibody prevalence rate against pertussis （PT） | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0]
  Antibody prevalence rate against pertussis （FHA） | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0]
  Antibody prevalence rate against tetanus toxin | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0]
  Antibody prevalence rate against polio virus serotype 1 | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0]
  Antibody prevalence rate against polio virus serotype 2 | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0]
  Antibody prevalence rate against polio virus serotype 3 | 100.0 [78.2 to 100.0] | 100.0 [78.2 to 100.0]

13. Secondary Outcome: Geometric Mean Antibody Titer Against Diphtheria Toxin
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310-High | BK1310-Low
Number analyzed (Participants) | 15 | 15
IU/mL | 12.9090 [8.0735 to 20.6406] | 10.2457 [6.2247 to 16.8642]

14. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis （PT）
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310-High | BK1310-Low
Number analyzed (Participants) | 15 | 15
EU/mL | 230.34 [167.63 to 316.52] | 223.85 [146.30 to 342.50]

15. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis （FHA）
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310-High | BK1310-Low
Number analyzed (Participants) | 15 | 15
EU/mL | 122.20 [73.26 to 203.83] | 85.52 [53.89 to 135.72]

16. Secondary Outcome: Geometric Mean Antibody Titer Against Tetanus Toxin
Time Frame: 4 weeks after the booster dose (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310-High | BK1310-Low
Number analyzed (Participants) | 15 | 15
IU/mL | 1.1670 [0.7576 to 1.7976] | 1.0640 [0.6375 to 1.7759]

17. Secondary Outcome: Fold Change in Geometric Mean Antibody Titer Against Polio Virus
Time Frame: Baseline and 4 weeks after the primary immunization (Visit 6)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | BK1310-High | BK1310-Low
Number analyzed (Participants) | 15 | 15
fold change
  Geometric mean antibody titer against polio virus serotype 1 | 4597.60 [2689.05 to 7860.76] | 1910.85 [1167.05 to 3128.69]
  Geometric mean antibody titer against polio virus serotype 2 | 7822.06 [5970.43 to 10247.94] | 6501.99 [4322.77 to 9779.82]
  Geometric mean antibody titer against polio virus serotype 3 | 4815.04 [3378.24 to 6862.93] | 4096.00 [2357.39 to 7116.87]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Arm/Group | BK1310-High | BK1310-Low | BK1310 | ActHIB® and Tetrabik (Control)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/171 | 0/169
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 8/171 | 5/169
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15 | 162/171 | 163/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BK1310-High (N=15) | BK1310-Low (N=15) | BK1310 (N=171) | ActHIB® and Tetrabik (Control) (N=169)
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 2
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Infantile haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Kawasaki's disease (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BK1310-High (N=15) | BK1310-Low (N=15) | BK1310 (N=171) | ActHIB® and Tetrabik (Control) (N=169)
Eye discharge (Eye disorders) | 0 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 4 | 5
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Crying (General disorders) | 4 | 1 | 45 | 41
Injection site erythema (General disorders) | 12 | 10 | 133 | 124
Injection site induration (General disorders) | 13 | 7 | 92 | 66
Injection site pain (General disorders) | 2 | 0 | 20 | 12
Injection site swelling (General disorders) | 9 | 4 | 60 | 55
Irritability postvaccinal (General disorders) | 2 | 2 | 27 | 17
Pyrexia (General disorders) | 10 | 9 | 114 | 104
Bronchitis (Infections and infestations) | 0 | 2 | 11 | 7
Conjunctivitis (Infections and infestations) | 0 | 1 | 4 | 8
Dermatitis infected (Infections and infestations) | 1 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 1 | 2 | 2
Gastroenteritis (Infections and infestations) | 1 | 2 | 4 | 4
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 4 | 4
Hordeolum (Infections and infestations) | 0 | 1 | 1 | 0
Impetigo (Infections and infestations) | 1 | 0 | 5 | 3
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 11 | 6 | 39 | 31
Otitis media acute (Infections and infestations) | 2 | 2 | 3 | 3
Pharyngitis (Infections and infestations) | 0 | 1 | 3 | 5
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 14 | 8
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 8 | 11
Viral rash (Infections and infestations) | 0 | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 19 | 19
Hypersomnia (Nervous system disorders) | 5 | 1 | 52 | 35
Insomnia (Psychiatric disorders) | 4 | 3 | 28 | 23
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 2 | 13 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2 | 15 | 5
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 3 | 9 | 8
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 9 | 10
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT02992925/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT02992925/SAP_001.pdf